CLINICAL TRIAL: NCT05908149
Title: Gait Analysis in Patients With Hemiplegia Using Insole Splint.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Avraam Ploumis, Director of Physical Medicine and Rehabilitation Clinic, University of Ioannina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10/12-4-2023 (T.34)
Record Dates: First submitted 2023-05-30; First posted 2023-06-18 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Gait, Hemiplegic; Splints; EMG
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HEMIPLEGIC PATIENTS (Experimental): HEMIPLEGIC PATIENTS WITH PES EQUINUS WILL BE EXAMINED BY GAIT ANALYSIS WITH AND WITHOUT THE INSOLE SPLINT, RANDOMLY
  Interventions: Device: Insole Splint

INTERVENTIONS:
Device: Insole Splint — Insole splint used in 'Pes equinus' in patients with hemiplegia

SUMMARY:
The goal of this clinical trial is to compare the gait of patients with hemiplegia, with or without the use of insole splint. The main questions it aims to answer are:

Does the insole splint improve the gait of these patients? Does any difference exist in the use of muscles?

Participants will have to walk in the gait analysis' aisle with and without the insole splint, using wireless EMG device.

ELIGIBILITY:
Inclusion Criteria:

* Patients that can walk with or without the splint, having their first stroke episode at least two months ago and their hospitalisation period does not overcome six months, having also a diagnosis from a neurologist coming with a Brain CT-scan.
* Patients must have use the insole splint during physiotherapy sessions for at least 1 week before their inclusion in the trial.
* Patients must be able to communicate and fully understand the instructions given by the researchers.
* Researchers are going to try to have a sex ratio 50/50.
* Patients' age is going to be between 18-70 years.
* Functional Ambulation Category: FAC > 2
* Modified Ashworth Scale of the affected lower Limb (MAS): MAS ≤2
* Normal Gait before the stroke.

Exclusion Criteria:

* Peripheral Neurological Damage.
* Past or ongoing orthopedic or reumatologic disease that bothers patient's gait.
* Past damage of the Central Nervous System.
* Dermatologic problems or human factors that limitate the use of insole splint.
* Patients must not have used intramuscular botox injection recently.
* Patients with low motivation and low perception are also excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gait speed | up to 6 months
  Patients are going to walk 15 metres with speed (meter/second) decided from the patient himself.
Gait cadence | up to 6 months
  Patients are going to walk 15 meters with speed decided from the patient himself and will measure cadence (number of full steps per minute)
Gait angles | up to 6 months
  Patients are going to walk 15 meters with speed decided from the patient himself. More specific, the investigators are going to count Ankle angles, Knee angles, Hip angles (in degrees) during gait.
Stride length | up to 6 months
  Patients are going to walk 15 meters with speed decided from the patient himself. More specific, the investigators are going to count Stride length (a full walking cycle of both feet making 1 step each)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Medicine and Rehabilitation, University Hospital of Ioannina, Ioannina, Greece